CLINICAL TRIAL: NCT05839873
Title: Abbott Ventricular Tachycardia Post Approval Study
Brief Title: Abbott Ventricular Tachycardia PAS
Status: Active, not recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10471
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Treatment Group: Single Arm Group to receive ablation.
  Interventions: Device: FlexAbility SE Ablation Catheter

INTERVENTIONS:
Device: FlexAbility SE Ablation Catheter — Subjects receive ablation treatment.

SUMMARY:
This post-approval study (PAS) is designed to provide continued clinical evidence to confirm the long-term safety and effectiveness of the FlexAbilityTM Ablation Catheter, Sensor EnabledTM (FlexAbility SE) for the treatment of ventricular tachycardia in a post-market environment. This is a prospective, single arm, open-label, multi-center, observational study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legally acceptable representative or parent/guardian (as applicable) must provide written informed consent prior to any clinical investigation-related procedure
2. Subjects who have recurrent, drug-refractory, sustained MMVT with non-ischemic structural heart disease and a clinical decision has been made to use FlexAbility SE for an ablation procedure prior to enrollment in the research study
3. Refractory (i.e. not effective, not tolerated or not desired) to at least one Class I/III anti-arrhythmic medication for treatment of MMVT
4. Implanted with a market released ICD or CRT-D prior to the Index Ablation Procedure
5. Able and willing to comply with all study requirements

Exclusion Criteria:

1. Documented or known intracardiac thrombus or myxoma
2. Active systemic infection
3. History of atriotomy or ventriculotomy within 4 weeks prior to the Index Ablation Procedure
4. Patients with prosthetic valves as the catheter may damage the prosthesis
5. Unable to receive heparin or an acceptable alternative to achieve adequate anticoagulation

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This clinical investigation will enroll subjects of all genders who have recurrent, drug-refractory, sustained monomorphic ventricular tachycardia in patients with non-ischemic structural heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Rate of study device- and/or Study Ablation Procedure-related SAEs through 12 months post Index Ablation Procedure. | 12 Month
Composite of 12-month freedom from VT recurrence, death, and cardiac transplantation | 12 Month

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Ruffner, PhD, Study Director — Clinical Program Director
Locations (11):
- United States (11):
  - NCH Healthcare System, Naples, Florida
  - St. Vincent Hospital, Indianapolis, Indiana
  - Kansas City Cardiac Arrhythmia Research Foundation, Overland Park, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - VA Medical Center Minneapolis, Minneapolis, Minnesota
  - Carolinas Medical Center, Charlotte, North Carolina
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt Heart & Vascular Institute, Nashville, Tennessee
  - Baylor Scott & White Heart & Vascular Hospital, Dallas, Texas
  - University of Utah Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No